CLINICAL TRIAL: NCT05781464
Title: Effect of Prolonged Slow Expiration Technique on Blood Gases Among Neonates With Pneumonia
Brief Title: Effect of Prolonged Slow Expiration Technique on Blood Gases Among Pneumatic Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moshira Mohamed Metwally, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NoP.T.REC/012/003676
Record Dates: First submitted 2023-02-26; First posted 2023-03-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Drainage, Postural; Vibration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional chest physiotherapy (Placebo Comparator): This group receives traditional chest physiotherapy that include postural drainage, percussion and vibration ( manually or by a vibrator) in each session which is twice daily from admission to neonatal intensive care unit till discharge
  Interventions: Procedure: Traditional chest physiotherapy
- Prolonged slow expiration technique and traditional chest physiotherapy (Active Comparator): This group receives traditional chest physiotherapy that include postural drainage, percussion and vibration ( manually or by a vibrator) plus prolonged slow expiration technique in each session which is twice daily from admission in neonatal intensive care unit till discharge.
  Interventions: Procedure: Traditional chest physiotherapy; Procedure: Prolonged slow expiration technique

INTERVENTIONS:
Procedure: Traditional chest physiotherapy — Postural drainage: the patient is positioned in postural drainage so that gravity had the maximum effect on the lung segment that needed to be drained, all lung zones are emphasised in positional initiatives for babies.
  Percussion is the rhythmic striking of the chest wall with cupped hands for 1 to 2 minutes at a time.
  Vibration is performed by placing fingers on the chest wall over the segment being drained and isometrically contracting the forearm and hand muscles to produce a vibratory motion.
  Vibration is accomplished either through manual vibratory motion of the therapist's fingers on the infant's chest wall or through the use of a mechanical vibrator ( Foreo vibrator).
  Other Names: Postural drainage; Percussion; Vibration; Foreo Vibrator
Procedure: Prolonged slow expiration technique — The therapist places one hand on the thorax below the suprasternal notch and the other hand over the upper abdomen while the neonate is supine. Both hands will have hypothenar contact with the thorax and abdomen. At the end of the expiratory phase, the therapist places a compression force with both hands. Compression at the end of expiration with hypothenar eminence is kept for 2 or 3 breathing cycles. This technique is repeated several times, with a rest time between applications of about 5 or 10 spontaneous breaths.
  Arms: Prolonged slow expiration technique and traditional chest physiotherapy

SUMMARY:
Pneumonia is a medical condition that, if not treated promptly, can lead to life- threatening complications. The prolonged slow expiration technique is a new type of chest physiotherapy that helps infants discharge bronchial secretions which accumulated due to pneumonia.

DETAILED DESCRIPTION:
Pneumonia is an infective lung condition that is one of the most common risk factors for neonatal death. Pulmonary infections, most common caused by anaerobic bacterial infection, result in the accumulation of pus in the pleural cavity. Preterms, neonates with respiratory infections, and underdeveloped lungs all require the use of a prolonged slow expiration technique.

Prolonged slow expiration technique is the only chest clearance technique that provides both effective clearance and a soothing effect. Another recommendation for this technique is lack of application of emerging techniques of respiratory physiotherapy. Although the technique is effective, it is rarely in practice over the conventional methods of chest physiotherapy.

During prolonged slow expiration, intrathoracic pressure gradually rises due to thoracoabdominal compression, preventing bronchial collapse and flow disruption that occurs during forced expirations.

ELIGIBILITY:
Inclusion Criteria:

* Age since birth till 2 months
* Clinical findings of pneumonia: tachypnea, chest recession, fever, cyanosis and cough
* Radiological diagnosis of pneumonia (x-ray): lober or segmental consolidation, nodular or coarse patchy infiltration, diffuse haziness and air bronchogram.
* Neonates on oxygen therapy.

Exclusion Criteria:

* Neonates with congenital cardiopathy.
* Neonates with surgical incision in thorax or abdomen.
* Neonates with neurological intervention.
* Neonates with obstruction of upper air way.
* Neonates with gastroesophageal reflux and laryngeal affection.

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Change in arterial oxygen saturation (Sao2) | Change from Baseline SaO2 at 9 days
  Arterial oxygen saturation is assessed by standardized international monitor and measured by %
Change in systolic and diastolic blood pressure | Change from baseline systolic and diastolic blood pressure at 9 days
  Systolic and diastolic blood pressure are assessed by standardized international monitor and measured by millimeters of mercury ( mmHg)
Change in heart rate (HR) | Change from baseline HR at 9 days
  Heart rate is assessed by standardized international monitor and measured by beats per minute (BPM)
Change in temperature | Change from baseline temperature at 9 days
  Temperature is assessed by thermometer and measured by degree(°)
Change in power of hydrogen (PH) | Change from baseline PH at 9 days
  PH is assessed by blood gases machine and it is a scale used to specify the acidity or basicity of blood
Change in partial pressure of carbon dioxide (PaCO2) | Change from baseline PaCO2 at 9 days
  PaCO2 is assessed by blood gases machine and measured by mmHg and it serves as a marker of sufficient alveolar ventilation within the lungs
Change in bicarbonate (HCO3) | Change from baseline HCO3 at 9 days
  HCO3 is assessed by blood gases machine and measured by milliequivalents per litre (mEq/L) and it is used to detect electrolyte imbalance

CONTACTS AND LOCATIONS:
Overall Officials: Elham Salem, Study Chair — Cairo University
Locations (1):
- Faculty of physical Therapy, Giza, Egypt

REFERENCES:
- [Background] Lievens L, Vandenplas Y, Vanlaethem S, Van Ginderdeuren F. Prolonged Slow Expiration Technique and Gastroesophageal Reflux in Infants Under the Age of 1 Year. Front Pediatr. 2021 Sep 8;9:722452. doi: 10.3389/fped.2021.722452. eCollection 2021. PMID 34568241
- [Background] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404